CLINICAL TRIAL: NCT04134988
Title: Effects of an Adapted Physical Activity With an Interactive Gaming Platform on Fall Apprehension and Risk: A Randomized Controlled Trial
Brief Title: Effects of an Adapted Physical Activity With an Interactive Gaming Platform on Fear of Falling and Risk of Falling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Joel Belmin (Other)
Responsible Party: Sponsor-Investigator, Joel Belmin, Professor, RIVAGES
Organization: RIVAGES (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEDIMOOV_01
Record Dates: First submitted 2019-10-11; First posted 2019-10-22 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Falls (Accidents) in Old Age
Keywords: Fall; Older adults; Fear of falling; Serious games; Technology; Randomized controlled trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medimoov (Experimental): Bi-weekly 35-minute sessions of an adaptated physical activity administered by a psychomotor therapist for 8 weeks.
  Interventions: Other: Medimoov
- Standard rehabilitation (Active Comparator): Bi-weekly 35-minute sessions of the standard psychomotor therapy for 8 weeks.
  Interventions: Other: Standard psychomotor therapy

INTERVENTIONS:
Other: Medimoov — The Medimoov game platform (created by NaturalPad©) is a physio-gaming medical device, which comes in the form of functional and postural rehabilitation software. Associating movement capture and videogames, Medimoov contributes to the older adults' motivation and engagement and offers adapted physical activities.
  Arms: Medimoov
Other: Standard psychomotor therapy — Psychomotor therapists are among the professionals recommended by the French national health authority. They intervene on psychomotor dimensions of falls, namely the motor, sensory and cognitive aspects.
  Arms: Standard rehabilitation

SUMMARY:
This study evaluates the effects of an adapted physical activity with an interactive gaming platform on fall apprehension and risks. Half of the participants will receive a rehabilitation program using the Medimoov gaming program, the other half will receive the standard rehabilitation program.

DETAILED DESCRIPTION:
Medimoov is an innovative interactive gaming platform offering adapted physical activity. Like most serious games, it targets both physical and cognitive components. Studies that evaluate serious games lack an appropriate control group, thus this study aims to evaluate the efficacy of serious games played with the Medimoov platform on fear of falling and fall risks. This pilot study is an open randomized controlled trial in parallel groups with blind data collection for the primary outcome.

The intervention group will follow bi-weekly sessions with Medimoov. The control group will follow the usual rehabilitation program: the standard psychomotor therapy program.

Both interventions will be consistent with rehabilitation programs prescribed by participants' physicians. Each intervention, guided by a psychomotor therapist, will last eight weeks with bi-weekly sessions of 35 minutes.

Participants will be randomly assigned to one of the two groups. Three assessments will be conducted focusing on physical and cognitive capacities. The first assessment will be conducted five or fewer days before the beginning of the rehabilitation program, the second will occur during week 4 and the third one during week 8, at the end of the rehabilitation program. Assessments will be blinded: assessors will not know the assigned group of each participant.

ELIGIBILITY:
Inclusion Criteria:

* To be at least 65 years old,
* To be able to give consent,
* French-speaking,
* To be able to stand upright in a bipedal position, feet together for a time greater than 10 seconds with/without an assistive device,
* To have a score ≥13 on the Short Fall Efficacy Scale (FES-I) (moderate fear of falling).

Exclusion Criteria:

* Not being able to answer the questionnaires,
* Not being able to correctly distinguish the elements on the screen,
* To be in palliative care,
* To be under a legal protection measure,
* To score under 16 at the Mini Mental State Examination,
* To have an acute pathology,
* To have had recent hip surgery (<2 months).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Change in the Score Physical Performance Battery | Before, at mid-term (Week 4) and at the end of the program (Week 8).
  This 5-minute test focuses on the static balance, walks, lower limb strength and fall risk. The score varies between 0 and 12, a score under 6 indicates a low performance and a high fall risk. Higher scores mean a better outcome.
Change in the Fall Efficacy Scale-International (FES-I) | Before, at mid-term (Week 4) and at the end of the program (Week 8).
  This five-minute questionnaire is composed of seven questions on daily activities and focus on the fear of falling. Each question can be scored between 1 (" Not at all concerned ") to 4 points (" Very concerned "). Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change in the Victoria Stroop test | Before, at mid-term (Week 4) and at the end of the program (Week 8)
  This 5-minute test to evaluate inhibition and selective attention is scored according to the realization time and errors in realization. The test includes three parts, the time of realization and the number or error are compared to a standard for each part of the test. Higher scores mean a worse outcome.
Change in the Trail Making Test A and B | Before, at mid-term (Week 4) and at the end of the program (Week 8)
  This evaluation focuses on executive functions including number and letter recognition, cognitive flexibility, visual scan, and motor functions. This evaluation lasts 10 minutes. The score of each test (A and B) is the number of seconds required to complete the task and is compared to a standard: for the Test A a score above 78 indicates a deficiency, for the Test B a score above 273 indicates a deficiency. Higher scores mean a worse outcome.
Change in the Timed Up And Go | Before, at mid-term (Week 4) and at the end of the program (Week 8)
  This test consists in standing up from a chair with armrest, walking three meters, turning around and coming back to sit. The test lasts less than one minute, fall risk is identified if the score is inferior than one and the duration of the test superior to 20 seconds.
Change in the One-Leg Stand test | Before, at mid-term (Week 4) and at the end of the program (Week 8)
  Standing in one leg as long as possible on each foot. This time is compared to a standard. Higher scores mean a better outcome.
Satisfaction questionnaire | At the end of the program (Week 8)
  Composed of 10 questions, its aim is to evaluate the participants' experience and the self-confidence after the rehabilitation program. The questionnaire lasts approximately 2 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Joël Belmin, MD, PhD, Principal Investigator — RIVAGES
Locations (1):
- Hôpitaux Universitaires Pitié Salpêtrière - Charles Foix et Sorbonne Université, Ivry-sur-Seine, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dargent-Molina P, Cassou B. Prévention des chutes chez les personnes âgées de plus de 75 ans vivant à leur domicile: analyse des interventions efficaces et perspectives de santé publique. Bull Épidémiologique Hebd. 2017;16-17:336-43.
- [Background] Tallon G, Seilles A, Melia G, et al. Intérêt du serious game Medimoov pour améliorer l'autonomie fonctionnelle chez la personne âgée institutionnalisée. Montpellier, 2015.
- [Background] Lister C, West JH, Cannon B, Sax T, Brodegard D. Just a fad? Gamification in health and fitness apps. JMIR Serious Games. 2014 Aug 4;2(2):e9. doi: 10.2196/games.3413. PMID 25654660
- [Background] Skjaeret N, Nawaz A, Morat T, Schoene D, Helbostad JL, Vereijken B. Exercise and rehabilitation delivered through exergames in older adults: An integrative review of technologies, safety and efficacy. Int J Med Inform. 2016 Jan;85(1):1-16. doi: 10.1016/j.ijmedinf.2015.10.008. Epub 2015 Oct 28. PMID 26559887
- [Background] Melia G, Seilles A, Tallon G. Évaluation d'un jeu sérieux thérapeutique. 2025; 4.
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Siegrist M. Test-Retest Reliability of Different Versions of the Stroop Test. J Psychol. 1997; 131: 299-306.
- [Background] Hauer KA, Kempen GI, Schwenk M, Yardley L, Beyer N, Todd C, Oster P, Zijlstra GA. Validity and sensitivity to change of the falls efficacy scales international to assess fear of falling in older adults with and without cognitive impairment. Gerontology. 2011;57(5):462-72. doi: 10.1159/000320054. Epub 2010 Oct 22. PMID 20975251
- [Background] Freire AN, Guerra RO, Alvarado B, Guralnik JM, Zunzunegui MV. Validity and reliability of the short physical performance battery in two diverse older adult populations in Quebec and Brazil. J Aging Health. 2012 Aug;24(5):863-78. doi: 10.1177/0898264312438551. Epub 2012 Mar 15. PMID 22422762
- [Background] Wagner S, Helmreich I, Dahmen N, Lieb K, Tadic A. Reliability of three alternate forms of the trail making tests a and B. Arch Clin Neuropsychol. 2011 Jun;26(4):314-21. doi: 10.1093/arclin/acr024. Epub 2011 May 15. PMID 21576092
- [Derived] Lapierre N, Um Din N, Igout M, Chevrier J, Belmin J. Effects of a Rehabilitation Program Using a Patient-Personalized Exergame on Fear of Falling and Risk of Falls in Vulnerable Older Adults: Protocol for a Randomized Controlled Group Study. JMIR Res Protoc. 2021 Aug 26;10(8):e24665. doi: 10.2196/24665. PMID 34435968